CLINICAL TRIAL: NCT00204516
Title: Pilot Study of Intradermal Vaccination of Melanoma Patients With a Fixed Combination of mRNAs Compared to an Individualized Selection After Analysis of Antigen Expression in Tumor Tissue
Brief Title: Vaccination With Tumor mRNA in Metastatic Melanoma - Fixed Combination Versus Individual Selection of Targeted Antigens
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Thomas Eigentler, Study Coordinator, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNA-Mel-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Malignant Melanoma
Keywords: vaccination; mRNA
MeSH Terms: conditions — Melanoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (1):
- mRNA Vacc (Experimental)
  Interventions: Biological: mRNA coding for melanoma associated antigens; Drug: GM-CSF

INTERVENTIONS:
Biological: mRNA coding for melanoma associated antigens — mRNA vaccine s.c. applied weekly
Drug: GM-CSF — Given s.c. as adjuvant drug one day after vaccine

SUMMARY:
The purpose of the vaccination protocol is to induce specific immune responses against melanoma associated antigens by intradermal injections of mRNA coding for the corresponding antigen.

DETAILED DESCRIPTION:
vaccination protocol to induce clinically specific immune responses against melanoma associated antigens by intradermal injections of mRNA coding for the corresponding antigens. Half of patients is treated with mRNA coding for Melan-A, Mage-A1, Mage-A3, Survivin, GP100 and Tyrosinase. The other half of patients is treated with an individualized selection of mRNAs after analysis of overexpressed melanoma antigens in autologous tumor tissue. GM-CSF is used as an adjuvants. Phase I/II clinical trial to analyse safety and immune responses in stage III/IV melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* malignant melanoma stage III/IV
* fresh frozen tumor tissue available
* informed consent given
* Karnofsky >= 70%

Exclusion Criteria:

* brain metastasis
* parallel chemotherapy
* systemic treatment with glucocorticoids
* other malignancies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-04; Primary Completion 2011-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Tolerability | every 4 weeks
  Side effects will be monitored using CTCAE criteria. Tolerability and toxicity profiles will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, Prof. Dr., Principal Investigator — University of Tuebingen, Department of Dermatology
Locations (1):
- Department of Dermatology, University of Tuebingen, Tübingen, Germany